CLINICAL TRIAL: NCT04980365
Title: Psychology Mobile Apps for Parents in a Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sam Houston State University (Other)
Responsible Party: Principal Investigator, Chelsea Ratcliff, Assistant Professor, Sam Houston State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-2020-230
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Stress, Psychological
Keywords: Parental stress; Health Psychology; Mental health apps; Mindfulness; Gratitude
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Potential participants will be provided access to an informed consent form and baseline survey via Qualtrics. After baseline is completed and eligibility confirmed, the study coordinator will randomly assign the participant to one of three app-based intervention conditions: Gratitude, Mindfulness, or control group. Next, the study coordinator will email them to schedule a Zoom meeting. The meeting will last 15 minutes and participants will be informed of what app they will use. After a 14-day period, the study coordinator will send participants a follow-up survey, and a final follow-up Qualtrics survey one month after the intervention ends. Participants will receive $5 for completing the baseline questionnaire, $5 for the immediate post-survey, and $10 for the one-month follow-up survey (participants can receive up to $20). Participants recruited via PeRP will receive one credit for completing the baseline questionnaire, two for the post-survey, and one for the follow-up.
Who Masked: Participant
Masking Description: Participants will have knowledge of the intervention they will receive but will have no knowledge of the other interventions used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (Experimental): Participants will be asked to use the app Mindfulness Coach 10 minutes for 14 days.
  Interventions: Behavioral: Mindfulness
- Gratitude (Experimental): Participants will be asked to use the app Grateful 10 minutes for 14 days.
  Interventions: Behavioral: Gratitude
- Control (Active Comparator): Participants will be asked to use the app Day One daily for 10 minutes. Participants will be writing a daily journal entry describing what they ate during the previous day for 14 days.
  Interventions: Behavioral: Food Journal

INTERVENTIONS:
Behavioral: Mindfulness — Participants will be asked to use the app Mindfulness Coach daily for 10 minutes. Participants will follow app instructions for brief guided meditation sessions for 14 days.
  Arms: Mindfulness
Behavioral: Gratitude — Participants will be asked to use the app Grateful daily for 10 minutes. Participants will follow app instructions and will be answering to prompts related to gratitude provided by the app daily, for 10 minutes for 14 days.
  Arms: Gratitude
Behavioral: Food Journal — Participants will be asked to use the app Day One daily for 10 minutes. Participants will be writing a daily journal entry describing what they ate during the previous day for 14 days.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether parents of young children (aged 10 and under) think it is feasible (in other words, doable) and acceptable (in other words, satisfactory) to use a mobile app designed to provide personalized education and enrichment for 10 minutes/day for 14 days. The investigators hope to learn if it is reasonable to ask parents to use one of three different apps and if parents are satisfied with their participation in the study. If so, the investigators can continue to study the effect of these apps on parents' stress in future research.

The investigators also plan to evaluate the effect of these app-based interventions in lowering levels of stress in parents during the COVID-19 pandemic. By conducting this study, the investigators hope to learn if there are specific app-based interventions that will lead to a reduction in stress in parents, improved parental life satisfaction, and improved parent-child interactions. If the results of this study suggest these apps may be promising at reducing stress among parents, the investigators will continue doing research on these app-based interventions.

DETAILED DESCRIPTION:
Parents will be invited to participate in a research study to see what parents of young children (aged 10 and under) think of using one of three different mobile app-based interventions to improve parental life satisfaction. The study will be conducted by Dr. Chelsea Ratcliff and Dr. Hillary Langley, Assistant Professors of Psychology at Sam Houston State University. In addition to learning about parents' satisfaction with these app-based interventions, the investigators also plan to compare the effect of these app-based interventions on levels of parental stress, and on quality of parent-child interactions during the COVID-19 pandemic.

The purpose of this research is to learn if it is reasonable to ask parents to use one of three different apps and if parents are satisfied with their participation in the study. If so, the investigators can continue to study the effect of these apps. The investigators also plan to evaluate the effect of these app-based interventions in lowering levels of stress in parents. By conducting this study, the investigators hope to learn if there are specific app-based interventions that will lead to a reduction in stress in parents, improved parental life satisfaction, and improved parent-child interactions.

In order to be eligible to participate, participants must be 18 years old or older, and a parent or primary caregiver of a child/children aged 10 years or young. Participants will first consent to participate by signing their name electronically using the mouse at the end of this consent form and providing their name and email address so the investigators can maintain contact. After reading this consent form and agreeing to it, participants will be directed to complete the first survey, which will take about 30 minutes to complete. They will be asked to complete two short questionnaires to determine their eligibility for the study. Participants will receive a $5 gift card for completing the first questionnaire.

After completing the pre-intervention survey, participants will be randomly assigned to use one of three psychology mobile apps. The study coordinator will email them to set up a 15-minute Zoom meeting in order to provide more information about the intervention and to help download the app that they were assigned. After the 14-day period, the study coordinator will email participants a link to a 20-minute follow-up survey, and they will receive a $5 gift card for completing this survey. One month later, the study coordinator will email participants a link to the final follow-up survey, and you will receive a $10 gift card for completing this survey. Thus, participants can earn up to $20 in Amazon gift cards for participating in this study ($5 for the pre-intervention survey, $5 for the immediate post-intervention survey, and $10 for the one-month post-intervention survey).

ELIGIBILITY:
Inclusion Criteria:

1. Only individuals aged 18 and older will be allowed to participate in the current research (assessed by participant self-report).
2. Individuals must identify oneself as a parent or primary caregiver of a child/children aged 10 or under (assessed by participant self-report).
3. Participants who score 30 or higher in the Parent Stress Scale (PSS) measure.
4. Participants who reside in the U.S. and can understand and answer surveys in English.

Exclusion Criteria:

1. Individuals under 18
2. Non-English-speaking individuals
3. Individuals who do not consent to the survey.
4. Individuals who do not identify oneself as a parent or primary caregiver of a child/children under the age of 10 (assessed by participant self-report).
5. Individuals who score 30 or lower in the PSS measure.
6. Individuals who do not reside in the U.S.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Parental Stress Scale Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Parental stress will be measured with The Parental Stress Scale, an 18-item self report scale; scores range from 18-90.

SECONDARY OUTCOMES:
Five Facet Questionnaire: Short Form Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Trait mindfulness will be measured with the Five Facet Questionnaire: Short Form, a 15-item self-report scale; scores range from 15-75.
Gratitude Questionnaire-6 Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Trait gratitude will be measured with the Gratitude Questionnaire-6 (GQ-6), a 6-item self-report measure that ranges from 6-42.
Gratitude Resentment and Appreciation Test-Revised Short Form Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Trait gratitude will be measured with Gratitude Resentment and Appreciation Test-Revised Short Form (GRAT-R-SF), a 16-item self-report measure with scores ranging from 16-144.
Dyadic Adjustment Scale Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Perceptions of one's relationship with an intimate partner will be measured via the Dyadic Adjustment Scale (DAS-7), a 7-item self-report measure with scores ranging from 0-36.
Positive & Negative Affect Scores | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Positive and negative affect will be measured using the Positive and Negative Affect Schedule (PANAS), a 20-item self-report measure with PA scores ranging from 0-50 and NA scores ranging from 0-50.
Child-Parent Relationship Scale Closeness & Conflict Scores | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Parents' views of their relationship with their child will be measured with the Child-Parent Relationship Scale, a 15-item self-report measure, with 7 items assessing closeness (range 7-35) and 8 items assessing conflict (range 8-40).
Perceived Stress Scale Total Score | T1 (before intervention); T2 (immediately after intervention); T3 (1-month after intervention)
  Perceived stress will be measuring using the Perceived Stress Scale (PSS), a 10-item self-report measure with scores ranging from 0-40.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea G Ratcliff, Ph.D., Principal Investigator — Sam Houston State University
Locations (1):
- Sam Houston State University, Huntsville, Texas, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data with other researchers.

REFERENCES:
- [Derived] Ratcliff CG, Langley HA, Torres D, Anderson KS. Randomized controlled trial of brief app-based gratitude and mindfulness interventions for parents of young children. J Fam Psychol. 2025 Sep;39(6):848-860. doi: 10.1037/fam0001347. Epub 2025 Jun 9. PMID 40489175